CLINICAL TRIAL: NCT00003280
Title: A Randomized, Phase III Trial to Determine the Effect of Consolidation With Rituximab (IDEC C2B8-Mabthera) in Patients With CD20+ Follicular or Mantle Cell Lymphoma Having Received Induction Therapy With Rituximab Weekly x 4
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Follicular or Mantle Cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 35/98; SWS-SAKK-35/98; ICR-35/98; EU-98009
Record Dates: First submitted 1999-11-01; First posted 2003-09-24 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Lymphoma
Keywords: stage I mantle cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Rituximab

INTERVENTIONS:
Biological: rituximab

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. It is not yet known which treatment regimen is more effective for lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of different regimens of rituximab in treating patients who have follicular or mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the clinical efficacy of consolidation treatment with rituximab in terms of response rate in patients with follicular (closed to accrual 9/18/00) or mantle cell lymphoma.
* Compare the event free survival of patients after induction with or without consolidation.
* Compare the tolerability of these two treatment regimens by these patients.

OUTLINE: This is a randomized, open label, multicenter study. Patients are stratified according to participating center, histology (follicular (closed to accrual 9/18/00) vs mantle cell), status of disease (de novo vs relapsed vs resistant), response after induction (stable disease vs partial or complete response), and treatment status (treated vs untreated).

All patients receive induction therapy consisting of rituximab IV over 3-5 hours once a week during weeks 1-4. Patients are then randomized to one of two treatment arms.

* Arm I: Patients are observed.
* Arm II: Patients receive rituximab IV over 3-5 hours once a week during weeks 12, 20, 28, and 36.

Patients are followed weekly for the first month; every 8 weeks for the next 8 months; then at 12, 18, and 24 months; and then annually for the next 3 years.

PROJECTED ACCRUAL: A total of 240 patients (120 per arm) will be accrued for this study within 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven CD20 positive follicular (closed to accrual 9/18/00) or mantle cell lymphoma

  * Untreated "de novo" disease OR
  * Chemotherapy resistant disease OR
  * Relapsing disease
* Bidimensionally measurable disease
* No symptomatic CNS disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* No hepatitis B or C

Renal:

* Creatinine no greater than 2 times ULN

Cardiovascular:

* Ejection fraction at least 50%

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active opportunistic infections
* HIV negative
* No prior malignancy within 5 years except adequately treated carcinoma in situ of the cervix or localized nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior antibody based therapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (at least 6 weeks since nitrosoureas) and recovered
* No concurrent chemotherapy

Endocrine therapy:

* At least 4 weeks since prior corticosteroids, unless chronic dose no greater than 20 mg/day for nonlymphoma related condition
* No other concurrent corticosteroids

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 1998-01; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Ghielmini, MD, Study Chair — Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni
Locations (10):
- Switzerland (10):
  - Kantonspital Aarau, Aarau
  - Office of Walter Weber-Stadelman, Basel
  - University Hospital, Basel
  - Ospedale San Giovanni, Bellinzona
  - Inselspital, Bern, Bern
  - Hopital Cantonal Universitaire de Geneva, Geneva
  - Istituto Oncologico della Svizzera Italiana, Lugano
  - Burgerspital, Solothurn, Solothurn
  - City Hospital Triemli, Zurich
  - Klinik Hirslanden, Zurich

REFERENCES:
- [Result] Martinelli G, Schmitz SF, Utiger U, Cerny T, Hess U, Bassi S, Okkinga E, Stupp R, Stahel R, Heizmann M, Vorobiof D, Lohri A, Dietrich PY, Zucca E, Ghielmini M. Long-term follow-up of patients with follicular lymphoma receiving single-agent rituximab at two different schedules in trial SAKK 35/98. J Clin Oncol. 2010 Oct 10;28(29):4480-4. doi: 10.1200/JCO.2010.28.4786. Epub 2010 Aug 9. PMID 20697092
- [Result] Ghielmini M, Rufibach K, Salles G, Leoncini-Franscini L, Leger-Falandry C, Cogliatti S, Fey M, Martinelli G, Stahel R, Lohri A, Ketterer N, Wernli M, Cerny T, Schmitz SF. Single agent rituximab in patients with follicular or mantle cell lymphoma: clinical and biological factors that are predictive of response and event-free survival as well as the effect of rituximab on the immune system: a study of the Swiss Group for Clinical Cancer Research (SAKK). Ann Oncol. 2005 Oct;16(10):1675-82. doi: 10.1093/annonc/mdi320. Epub 2005 Jul 19. PMID 16030029
- [Result] Ghielmini M, Schmitz SF, Cogliatti S, Bertoni F, Waltzer U, Fey MF, Betticher DC, Schefer H, Pichert G, Stahel R, Ketterer N, Bargetzi M, Cerny T; Swiss Group for Clinical Cancer Research. Effect of single-agent rituximab given at the standard schedule or as prolonged treatment in patients with mantle cell lymphoma: a study of the Swiss Group for Clinical Cancer Research (SAKK). J Clin Oncol. 2005 Feb 1;23(4):705-11. doi: 10.1200/JCO.2005.04.164. Epub 2004 Dec 14. PMID 15598978
- [Result] Lee CS, Ashton-Key M, Cogliatti S, Rondeau S, Schmitz SF, Ghielmini M, Cragg MS, Johnson P. Expression of the inhibitory Fc gamma receptor IIB (FCGR2B, CD32B) on follicular lymphoma cells lowers the response rate to rituximab monotherapy (SAKK 35/98). Br J Haematol. 2015 Jan;168(1):145-8. doi: 10.1111/bjh.13071. Epub 2014 Aug 21. No abstract available. PMID 25142001